CLINICAL TRIAL: NCT00173082
Title: Metabolic Syndrome and Insulin Resistance in Primary Aldosteronism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700402
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; Insulin resistance; Metabolic syndrome; OGTT
MeSH Terms: conditions — Hyperaldosteronism; Insulin Resistance; Metabolic Syndrome | interventions — Glucose Tolerance Test

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Glucose tolerance test

SUMMARY:
Primary aldosteronism (PA) is occasionally associated with impaired glucose tolerance. Glucose intolerance, in general metabolic syndrome is caused by suppression of insulin release from the pancreas and suppression of insulin sensitivity of the target tissues. Several studies have suggested that impaired glucose tolerance in primary aldosteronism is due to an inability of the beta cells to release insulin by potassium depletion. It was suggested glucose intolerance in PA is caused by the suppression of insulin release related to hypopotassemia and compensatory increase of insulin sensitivity is observed in PA. The increased insulin secretory capacity associated with correction of negative potassium balance may account for the increase in plasma leptin after curing primary aldosteronism. The conclusion with respect to the possible causal relationship between diabetes mellitus (DM) and PA, however, can be obtained after the evaluation of the effect of surgical /pharmacological treatment of PA.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is occasionally associated with impaired glucose tolerance. Glucose intolerance, in general metabolic syndrome is caused by suppression of insulin release from the pancreas and suppression of insulin sensitivity of the target tissues. Several studies have suggested that impaired glucose tolerance in primary aldosteronism is due to an inability of the beta cells to release insulin by potassium depletion. It was suggested glucose intolerance in PA is caused by the suppression of insulin release related to hypopotassemia and compensatory increase of insulin sensitivity is observed in PA. The increased insulin secretory capacity associated with correction of negative potassium balance may account for the increase in plasma leptin after curing primary aldosteronism. The conclusion with respect to the possible causal relationship between DM and PA, however, can be obtained after the evaluation of the effect of surgical /pharmacological treatment of PA. From July 2005 to July 2008, patients with primary aldosteronism, hospitalized for a comprehensive study of the subtypes of primary aldosteronism before operation will receive informed consent about the insulin sensitivity test. In the present study, we measured insulin sensitivity via the ability to release insulin by the 75 g oral glucose tolerance test (OGTT) in PA to clarify the mechanisms of glucose intolerance in PA. Seventy-five gram OGTT was performed in PA before and after adrenalectomy. Within one minute, 75 g of glucose dissolved in 200 cc water was ingested. Venous blood samples were drawn at 0, 60, 120 minutes for determination of plasma glucose and plasma insulin levels. Serum potassium levels were measures at 0 minutes. Furthermore, the adipokines, HOMA, QUICKI, leptin, adiponectin, homocystine, C-reactive protein, proinflammatory cytokine and adhesion molecules were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Aldosteronism patients

Exclusion Criteria:

* Patients with pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-06; Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Study Chair — National Taiwan University Hospital; Vin-cent Wu, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Corry DB, Tuck ML. The effect of aldosterone on glucose metabolism. Curr Hypertens Rep. 2003 Apr;5(2):106-9. doi: 10.1007/s11906-003-0065-2. PMID 12642008
- [Background] Widimsky J Jr, Strauch B, Sindelka G, Skrha J. Can primary hyperaldosteronism be considered as a specific form of diabetes mellitus? Physiol Res. 2001;50(6):603-7. PMID 11829322
- [Background] Kreze A Sr, Kreze-Spirova E, Mikulecky M. Diabetes mellitus in primary aldosteronism. Bratisl Lek Listy. 2000;101(4):187-90. PMID 10914461